CLINICAL TRIAL: NCT05121233
Title: Local Anesthesia Versus Combined Local Anesthesia With Single Dose Analgesia on Pain Control During Thoracic Ultrasound Guided Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Ahmed AbdAllah, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: pain in TUS guided procedures
Record Dates: First submitted 2021-09-25; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Pleural Neoplasms; Aspiration, Respiratory; Pleural Effusion; Lung Neoplasms; Pneumothorax; Pyothorax
MeSH Terms: conditions — Pleural Neoplasms; Respiratory Aspiration; Pleural Effusion; Lung Neoplasms; Pneumothorax; Empyema, Pleural | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diclofenac (Active Comparator): Group A will receive a single dose 75 mg IV diclofenac by infusion prior to the procedure
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator): Group B who will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac — a single dose 75 mg IV diclofenac by infusion prior to the procedure
  Arms: Diclofenac
Drug: Placebo — single dose iv placebo (saline ) by infusion prior to the procedure
  Arms: Placebo

SUMMARY:
This study aims to evaluate the efficacy of single dose analgesia in combination with local anesthesia to control pain during Trans Ultrasound guided procedures. It also aims to assess the effect of its use on procedure performance time and rate of complications occurrence compared to local anesthesia alone.

DETAILED DESCRIPTION:
Interventional thoracic ultrasonography (TUS) includes both diagnostic and therapeutic procedures. Fine-needle aspiration biopsy , Tru-cut Pleural or lung parenchymal biopsy and Cope or Abrams needles pleural biopsies are examples of diagnostic procedures while ultrasound guided thoracentesis, pleural aspiration for pneumothorax, placement of chest tubes, and indwelling catheter insertion, or pleurodesis are common therapeutic procedures.

Thoracic ultrasound guided procedures are safe and tolerable. Pain, pneumothorax, bleeding, infection, and procedure failure are the possible complications of TUS guided procedures. Lidocaine 1% should be infiltrated prior to the procedure, paying particular attention to the skin, periosteum and the pleura as a local anesthesia.

To reduce pain, analgesia should be considered as premedication. Despite the apparent common sense of this approach, there is little established evidence of the effect from these medications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders.
* Patients with pleural effusion, pneumothorax, lung mass or chest wall mass accessible for thoracic ultrasound guided intervention

Exclusion Criteria:

* Children and patients less than 18 years old.
* Pregnant and lactating ladies.
* Patients with disturbed level of consciousness.
* Patients with known bleeding disorders.
* Patients with advanced liver and kidney disorders.
* Patients with known hypersensitivity to NSAIDS.
* Patients with chronic chest diseases.
* Patients who refuse to participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity assessed by Numerical Rating Scale (NRS) | 30 minutes
  evaluate the efficacy of single dose analgesia in combination with local anaesthesia to control pain during TUS guided procedures by Numerical Rating Scale , patient is asked to indicate his/her perceived pain intensity , the patient grades their own pain on a scale between 1 to 10
Satisfaction assessed by the Visual Analogue Scale (VAS) | 30 minutes
  satisfaction assessment by Visual Analogue Scale , series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable"
performance time of transthoracic ultrasound guided procedures | up to 20 minutes
  assess the effect of its use with local anaesthesia on procedure performance compared to local anaesthesia alone

REFERENCES:
- [Background] Almolla J, Balconi G. Interventional ultrasonography of the chest: Techniques and indications. J Ultrasound. 2011 Mar;14(1):28-36. doi: 10.1016/j.jus.2011.01.005. Epub 2011 Feb 12. PMID 23396954
- [Background] Havelock T, Teoh R, Laws D, Gleeson F; BTS Pleural Disease Guideline Group. Pleural procedures and thoracic ultrasound: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii61-76. doi: 10.1136/thx.2010.137026. No abstract available. PMID 20696688
- [Background] Rahman NM, Pepperell J, Rehal S, Saba T, Tang A, Ali N, West A, Hettiarachchi G, Mukherjee D, Samuel J, Bentley A, Dowson L, Miles J, Ryan CF, Yoneda KY, Chauhan A, Corcoran JP, Psallidas I, Wrightson JM, Hallifax R, Davies HE, Lee YC, Dobson M, Hedley EL, Seaton D, Russell N, Chapman M, McFadyen BM, Shaw RA, Davies RJ, Maskell NA, Nunn AJ, Miller RF. Effect of Opioids vs NSAIDs and Larger vs Smaller Chest Tube Size on Pain Control and Pleurodesis Efficacy Among Patients With Malignant Pleural Effusion: The TIME1 Randomized Clinical Trial. JAMA. 2015 Dec 22-29;314(24):2641-53. doi: 10.1001/jama.2015.16840. PMID 26720026
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510